CLINICAL TRIAL: NCT03410706
Title: Xarelto® for Real Life Anticoagulation in Pulmonary Embolism (PE) in China
Brief Title: Xarelto for Real Life Anticoagulation in Pulmonary Embolism (PE) in China
Acronym: XAPEC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18799
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Embolism
Keywords: Venous thromboembolism; Anticoagulation; Rivaroxaban; Observation study
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban: Anticoagulation with rivaroxaban
  Interventions: Drug: Rivaroxaban(Xarelto, BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban(Xarelto, BAY 59-7939) — The dosage and the anticoagulation duration is decided by investigators. As list in product information, the PE treatment dosage of rivaroxaban is 15mg bid for first 21 days and then 20mg qd. If CrCl is 30-49 ml/min and bleeding risk is over VTE recurrence risk, 20mg qd can be replaced with 15mg qd.

SUMMARY:
EINSTEIN PE study demonstrated that rivaroxaban is at least as effective as the current standard therapy with 51% relative risk reduction of major bleeding (1.1% vs. 2.2%, HR 0.49, 95% CI, 0.31-0.79), in the treatment and secondary prevention of PE. However these patients were required to meet strict eligibility criteria. Little is known about PE treatment in China in routine clinical practice and in a real world study patients at higher or lower risk for adverse events can possibly recruited. Bayer conducts this study to yield post-authorization safety information in rivaroxaban under real-life conditions in China.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, who are at >=18 years
* Diagnosis of acute symptomatic or asymptomatic PE, objectively confirmed
* Indication for anticoagulation therapy for at least 3 months (as assessed by the attending investigator)
* Willing to participate in this study, having given informed consent and willing to participate in the routine follow-up during the period of rivaroxaban treatment.

Exclusion Criteria:

* Pre-treatment with any anticoagulant for the index PE more than the 2 weeks.
* Patients with another indication for anticoagulation other than VTE.
* Patients who participated in another study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in Tertiary hospitals
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Major bleedings | Up to 12 months
  Major bleedings defined as overt bleeding associated with: A fall in hemoglobin of ≥2 g/dL; or a transfusion of ≥2 units of packed red blood cells or whole blood; or occurrence at a critical site: intracranial, intra-spinal, intraocular, pericardial, intra-articular, intra-muscular with compartment syndrome, retroperitoneal; or death.

SECONDARY OUTCOMES:
Symptomatic recurrent venous thromboembolic events | Up to 12 months
  Will be confirmed by objective diagnostic tools, such as compression ultrasound, venography, CT scan or ventilation/perfusion lung scan, according to the real clinical practice.
Major adverse cardiac events | Up to 12 months
  Including myocardial infarction and cardiac death
Other symptomatic thromboembolic events | Up to 12 months
  As defined by Standardized MedDRA Query 'Embolic and thrombotic events
Drug utilization | Up to 12 months
  Dosage, duration, discontinuation, reason for any drug switch or interruption, co-medications
Number of participants with adverse events and serious adverse events | Up to 12 months
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
  An AE is serious (SAE) if it:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization (see exceptions below)
  * Results in persistent or significant disability or incapacity
  * Is a congenital anomaly or birth defect
  * Is medically important.
Patient treatment satisfaction by using questionnaire of ACTS (Anti-Clot Treatment Scale) | Up to 12 months
  The Anti-Clot Treatment Scale (ACTS) is a 17-item patient-reported measure of satisfaction with anticoagulant treatment. It includes 13 items about the burdens and 4 items about the benefit of ACT.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/